CLINICAL TRIAL: NCT02838862
Title: Identification of Biomarker Profiles for Individualized Prognostic Stratification and Therapy in Patients With Gastroenteropancreatic Neuroendocrine Neoplasia (GEP-NEN)
Brief Title: Identification of Biomarker Profiles GEP-NEN Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Franck Billmann, Director Section for Endocrine Surgery, University Hospital Schleswig-Holstein
Other Study IDs: 16-087
Record Dates: First submitted 2016-07-16; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine Tumors; MALDI-MS; Proteomics; Biomarkers, Tumor; Precision Medicine
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — proteomic analysis (MALDI-MS) applied to existing pathology specimens of Neuroendocrine tumors (paraffin-embedded specimens, FFPE).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Response to Therapy
- No therapy response

SUMMARY:
Although gastroenteropancreatic neuroendocrine neoplasia (GEP-NEN) were considered for years as rare tumors, their incidences are increasing. Due to their potential of early metastases and their heterogenous response to therapy, these tumors are important clinical entities. A major problem remains the impossibility to adequately predict tumors' response to treatment, precluding an individualized therapy. Further, there is no method to efficiently screen these tumors. Protein based analyses (proteomic analyses) gain in interest as methods to address this problematic.

The present study was designed to investigate epidemiologic data of patients with GEP-NEN and to answer following questions using proteomic analysis applied to existing pathology specimens (paraffin-embedded specimens, FFPE): is it possible to explore protein signatures in this type of tumors? Is the response to therapy predictable using specific protein signatures? Is the tumor's tendency to metastasize related to specific protein signatures?

DETAILED DESCRIPTION:
Gastroenteropancreatic neuroendocrine neoplasia (GEP-NEN) were considered for years as rare tumors. In last years however, their incidences are increasing (3,65 / 100.000 / year) [Lawrence et al., 2011; Friling et al, 2014]. These tumors are important clinical entities: 1) 40-95% of tumors have metastasized at diagnosis, 2) evidence-based data dealing with the therapeutic strategy and screening are still scarce.

A central problem remains the impossibility to adequately predict the response to surgery, chemotherapy, radiochemotherapy, peptid-receptor-based Radiotherapy or biotherapy, precluding an individualized therapy (precision medicine) [Rinke et al., 2014]. An actual research topic in these patients is the identification of patient markers allowing an response prediction. Moreover, researchers try to identify tumor markers in patients with unknown primary in order to locate the origin of metastases. Further, identification of tumor specific markers would allow the development of screening strategies in GEP-NEN. Due to the ability of these techniques to describe the biological heterogenity of a tumor, proteomics (protein based analysis methods) are promising in the present problematic [Bezabeh et al., 2014; Löhr et al., 2006; Pan et al., 2013].

The present study was designed to investigate epidemiologic data of patients with GEP-NEN and to answer following questions using proteomic analysis (MALDI-MS) applied to existing pathology specimens (paraffin-embedded specimens, FFPE): is it possible to explore protein signatures in this type of tumors? Is the response to therapy predictable using specific protein signatures? Is the tumor's tendency to metastasize related to specific protein signatures? The present investigation explores the GEP-NEN database/register of following institutions: University Hospital Schleswig Holstein, University hospital of Freiburg, Agaplesion Hospital Rotenburg. The pathology specimens of the studied register-population, were identified in the biobank and pathology-institutes of the participating hospitals and investigated using MALDI-MS technique.

ELIGIBILITY:
Inclusion Criteria:

* GEP-NEN

Exclusion Criteria:

* Absence of histological confirmation of the diagnosis
* Absence of pathology specimen to evaluate using MALDI-MS

Ages: 12 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: GEP-NEN Patients registered in the institutional NEN Registries
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Response to Therapy (Surgery, Chemotherapy, Radiotherapy, etc.) | 12 months - 10 years (retrospective groups)

SECONDARY OUTCOMES:
Overall Survival | 12 months - 10 years (retrospective groups)
Disease free Survival | 12 months - 10 years (retrospective groups)
Morbidity | 12 months - 10 years (retrospective groups)
Mortality | 12 months - 10 years (retrospective groups)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Keck, MD, PhD, Study Chair — University Hospital Lübeck - Department of Surgery
Locations (3):
- Germany (3):
  - University Hospital Freiburg - Department of Surgery, Freiburg im Breisgau, Baden-Wurttemberg
  - University Hospital SH - Campus Lübeck - Department of Surgery, Lübeck, Schleswig-Holstein
  - Agaplesion Diakonieklinikum Rotenburg - Department of Surgery, Rotenburg (Wümme)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bezabeh T, Ijare OB, Nikulin AE, Somorjai RL, Smith IC. MRS-based Metabolomics in Cancer Research. Magn Reson Insights. 2014 Feb 13;7:1-14. doi: 10.4137/MRI.S13755. eCollection 2014. PMID 25114549
- [Background] Frilling A, Modlin IM, Kidd M, Russell C, Breitenstein S, Salem R, Kwekkeboom D, Lau WY, Klersy C, Vilgrain V, Davidson B, Siegler M, Caplin M, Solcia E, Schilsky R; Working Group on Neuroendocrine Liver Metastases. Recommendations for management of patients with neuroendocrine liver metastases. Lancet Oncol. 2014 Jan;15(1):e8-21. doi: 10.1016/S1470-2045(13)70362-0. PMID 24384494
- [Background] Lawrence B, Gustafsson BI, Chan A, Svejda B, Kidd M, Modlin IM. The epidemiology of gastroenteropancreatic neuroendocrine tumors. Endocrinol Metab Clin North Am. 2011 Mar;40(1):1-18, vii. doi: 10.1016/j.ecl.2010.12.005. PMID 21349409
- [Background] Lohr JM, Faissner R, Findeisen P, Neumaier M. [Proteome analysis--basis for individualized pancreatic carcinoma therapy?]. Internist (Berl). 2006 Jun;47 Suppl 1:S40-8. doi: 10.1007/s00108-006-1634-7. German. PMID 16773365
- [Background] Pan S, Brentnall TA, Kelly K, Chen R. Tissue proteomics in pancreatic cancer study: discovery, emerging technologies, and challenges. Proteomics. 2013 Feb;13(3-4):710-21. doi: 10.1002/pmic.201200319. Epub 2013 Jan 7. PMID 23125171
- [Background] Rinke A, Arnold R. Aktuelle Therapie neuroendokriner Tumoren. Arzneimitteltherapie 2014;32:2-13